CLINICAL TRIAL: NCT00733759
Title: The Evaluation of Intra-cardiac Shunts in Patients With Pulmonary Arteriovenous Malformations
Brief Title: Contrast Echocardiography in Patients With Pulmonary Arteriovenous Malformations (PAVMs)
Status: Withdrawn | Type: Observational
Why Stopped: Unable to recruit patients due to technical issues following submission
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: IC/CLS10
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Pulmonary Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Pulmonary arteriovenous malformations (PAVMs) are thin-walled abnormal vessels which provide direct capillary-free communications between the pulmonary and systemic circulations. Patients with PAVMs have usually have low blood oxygen levels and are at risk of other complications including strokes, brain abscesses, pregnancy-related complications and haemorrhage. We hypothesise that the complications of PAVM patients arise from their PAVMs and not the more recognised intracardiac forms of shunting. We propose to perform echocardiograms to enable assessment of the presence of other causes of capillary-free communications between the pulmonary and systemic circulations.

ELIGIBILITY:
Inclusion Criteria:

* patients with pulmonary arteriovenous malformations (PAVMs)

Exclusion Criteria:

* unable to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pulmonary arteriovneous malformations
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2004-02 (Estimated); Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire L Shovlin, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Hammersmith Campus, London, United Kingdom